CLINICAL TRIAL: NCT06515418
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm Proof-of-Concept Study to Investigate Efficacy and Safety of Oral Azelaprag Plus Once Weekly Tirzepatide Compared with Tirzepatide Alone in Participants with Obesity Aged 55 Years and Over (STRIDES)
Brief Title: Efficacy and Safety of Oral Azelaprag Plus Once Weekly Tirzepatide Compared with Tirzepatide Alone in Participants with Obesity Aged 55 Years and Over
Acronym: STRIDES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Dosing of both study drugs has been discontinued due to observation of liver transaminitis without clinically significant symptoms in some subjects receiving azelaprag. All participant visits have been completed.
Sponsor: BioAge Labs, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BGE-105-005
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Azelaprag; BGE-105; BioAge; Tirzepatide; Weight Management; GLP-1/GIP Receptor Agonist; STRIDES
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- A: Tirzepatide Monotherapy (Active Comparator): * Azelaprag placebo every morning
  * Azelaprag placebo every evening
  * Tirzepatide 5mg once weekly
  Interventions: Drug: Oral Placebo for Azelaprag (BGE-105); Drug: Tirzepatide
- B: Azelaprag once daily plus Tirzepatide (Experimental): * Azelaprag 300mg every morning
  * Azelaprag placebo every evening
  * Tirzepatide 5mg once weekly
  Interventions: Drug: Oral Azelaprag (BGE-105); Drug: Oral Placebo for Azelaprag (BGE-105); Drug: Tirzepatide
- C: Azelaprag twice daily plus Tirzepatide (Experimental): * Azelaprag 300mg every morning
  * Azelaprag 300mg every evening
  * Tirzepatide 5mg once weekly
  Interventions: Drug: Oral Azelaprag (BGE-105); Drug: Tirzepatide
- D: Azelaprag Monotherapy (Experimental): * Azelaprag 300mg every morning
  * Azelaprag 300mg every evening
  * Tirzepatide placebo once weekly
  Interventions: Drug: Oral Azelaprag (BGE-105); Drug: Tirzepatide Placebo

INTERVENTIONS:
Drug: Oral Azelaprag (BGE-105) — Capsules
  Other Names: BGE-105
  Arms: B: Azelaprag once daily plus Tirzepatide; C: Azelaprag twice daily plus Tirzepatide; D: Azelaprag Monotherapy
Drug: Oral Placebo for Azelaprag (BGE-105) — Capsules
  Other Names: Placebo
  Arms: A: Tirzepatide Monotherapy; B: Azelaprag once daily plus Tirzepatide
Drug: Tirzepatide — Subcutaneous Injection
  Arms: A: Tirzepatide Monotherapy; B: Azelaprag once daily plus Tirzepatide; C: Azelaprag twice daily plus Tirzepatide
Drug: Tirzepatide Placebo — Subcutaneous Injection
  Arms: D: Azelaprag Monotherapy

SUMMARY:
This study aims to find out how well a combination of oral azelaprag taken once a day (QD) or twice a day (BID), along with a weekly injection of tirzepatide, works for weight management in adults 55 years and older. The researchers are also looking at safety.

Estimated Study Length:

* with the optional prescreening, the study duration may be up to 48 weeks.
* the treatment duration will be 24 weeks followed by 12 weeks follow-up.
* the visit frequency will be every 2 weeks for the first 8 weeks of the treatment period and every 4 weeks thereafter.

DETAILED DESCRIPTION:
Clinical trial BGE-105-005 will determine if the addition of oral azelaprag to tirzepatide treatment will amplify overall weight loss in participants with obesity aged 55 years and older. BGE-105-005 is a randomized, double-blind, placebo-controlled, parallel-arm, multi-center study in approximately 220 adults ≥55 years old with body mass index (BMI) between 30 and 40 kg/m2 inclusive, at the time of screening. Participants will be randomly assigned to 1 of the 4 study arms (A-tirzepatide monotherapy, B-azelaprag 300 mg QD plus tirzepatide, C-azelaprag 300 mg BID plus tirzepatide, D-azelaprag 300 mg BID monotherapy). The primary endpoint will be the effect on body weight reduction as measured by mean percent change in body weight at 24 weeks in participants that received azelaprag plus tirzepatide versus tirzepatide alone. The study is intended to gather safety and efficacy data in the defined participant population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 55 years of age or older at the time of signing the informed consent.
2. Have a BMI between 30 and 40 kg/m2 inclusive at the time of screening.
3. Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

1. Have diagnosis of type 1 diabetes (T1D) or Type 2 diabetes (T2D) mellitus.
2. Have a self-reported change in body weight greater than 5 kg (11 lbs) within 90 days prior to screening.
3. Have a prior or planned surgical treatment or device-based therapy for obesity.
4. Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2).
5. Have an uncontrolled thyroid disease.
6. Have obesity induced by endocrinological disorders.
7. Have biopsy-confirmed nonalcoholic steatohepatitis (NASH), also known as metabolic dysfunction-associated steatohepatitis (MASH).
8. Have a known history or presence of severe active acute or chronic livers disease or acute or chronic pancreatitis, or exocrine pancreatic insufficiency.
9. Have a known history or presence of symptomatic gallbladder disease within the past 2 years.
10. Have a medically significant cardiovascular condition.
11. Have a history of active or untreated malignancy within the last 5 years.
12. Have a history of significant active or unstable major depressive disorder or other severe psychiatric disorder within the last 2 years.
13. Have any lifetime history of a suicide attempt.
14. Have a known clinically significant gastric emptying abnormality.
15. Have had previous or are currently on treatment with a GLP-1R agonist or tirzepatide (a dual agonist of GLP-1 and GIP receptors).
16. Are currently using warfarin.
17. Have used any weight loss drugs, including herbal or nutritional supplements, within 90 days of screening.
18. Have current or history of treatment with medications that may cause significant weight gain within 90 days of screening.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Mean Percent Change in Body Weight (Azelaprag Once per Day) | Week 24
  Mean percent change in body weight from baseline to Week 24 in the 300 mg azelaprag once per day (QD) plus tirzepatide arm compared to tirzepatide alone arm
Mean Percent Change in Body Weight (Azelaprag Twice per Day) | Week 24
  Mean percent change in body weight from baseline to Week 24 in the 300 mg azelaprag twice per day (BID) plus tirzepatide arm compared to tirzepatide alone arm

SECONDARY OUTCOMES:
≥5% Body Weight Reduction | Week 24
  Proportion of study participants at 24 weeks who achieve ≥5% body weight reduction from baseline for azelaprag plus tirzepatide compared to tirzepatide alone
≥10% Body Weight Reduction | Week 24
  Proportion of study participants at 24 weeks who achieve ≥10% body weight reduction from baseline for azelaprag plus tirzepatide compared to tirzepatide alone
≥15% Body Weight Reduction | Week 24
  Proportion of study participants at 24 weeks who achieve ≥15% body weight reduction from baseline for azelaprag plus tirzepatide compared to tirzepatide alone
≥20% Body Weight Reduction | Week 24
  Proportion of study participants at 24 weeks who achieve ≥20% body weight reduction from baseline for azelaprag plus tirzepatide compared to tirzepatide alone
Body Weight Change | Week 24
  Change from baseline in body weight (kg) at 24 weeks for azelaprag plus tirzepatide compared to tirzepatide alone
Waist Circumference Change | Week 24
  Change from baseline in in waist circumference (cm) at 24 weeks for azelaprag plus tirzepatide compared to tirzepatide alone
Serious Adverse Events | Up to Week 36
  The incidence of serious adverse events (SAEs)
Treatment Emergent Adverse Events | Up to Week 36
  The incidence of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Site 110, Mesa, Arizona
  - Site 107, Los Angeles, California
  - Site 103, Montclair, California
  - Site 105, Spring Valley, California
  - Site 100, Louisville, Kentucky
  - Site 101, Marrero, Louisiana
  - Site 112, Boston, Massachusetts
  - Site 111, Troy, Michigan
  - Site 113, City of Saint Peters, Missouri
  - Site 106, Butte, Montana
  - Site 109, Fargo, North Dakota
  - Site 108, Beachwood, Ohio
  - Site 102, Dallas, Texas
  - Site 104, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Zepbound™ USPI — https://www.accessdata.fda.gov/drugsatfda_docs/label/2024/217806s003lbl.pdf